CLINICAL TRIAL: NCT00701649
Title: A Double Blind, Randomized, Placebo Controlled, Parallel Group Phase IIa Study to Evaluate Safety and Tolerability, Pharmacodynamic Effects and Exploratory Efficacy of an Anti-Angiotensin II Vaccine (CYT006-AngQb) in Patients With Mild to Moderate Essential Hypertension
Brief Title: Study to Evaluate Safety and Tolerability, Pharmacodynamic Effects and Exploratory Efficacy of a Vaccine Against Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Prof. Dr. med. Jürg Nussberger, Hôpital Nestlé 6027, CHUV, CH-1011 Lausanne, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT006-AngQb 02; Eudract No. 2007-005843-93
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension
Keywords: mild essential hypertension; moderate essential hypertension
MeSH Terms: conditions — Hypertension | interventions — CYT006-AngQb

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: CYT006-AngQb
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CYT006-AngQb — s.c.
  Arms: 1
Biological: Placebo — s.c.
  Arms: 2

SUMMARY:
CYT006-AngQb is a vaccine that induces a B-cell mediated immune response characterized by the generation of specific antibodies (IgG and IgM) against Angiotensin II. The vaccine is administered by subcutaneous injection.

The objectives of the study are:

* To evaluate safety and tolerability of 5 s.c. injections of 300µg CYT006-AngQb with Alhydrogel™ in patients with mild to moderate essential hypertension (hypertension Grade I and II).
* To assess pharmacodynamic effects, i.e. anti-Ang II immune response and renin- angiotensin system (RAS) biomarkers.
* To explore the effect on blood pressure using ABPM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate essential hypertension (Grade I and Grade II) with mean sitting office SBP =140-179 mmHg and/or mean sitting office DBP = 90-109 mmHg on 2 consecutive visits (screening and V1).
* Daytime blood pressure above threshold for definition of hypertension in the screening ABPM measurement (SBP >135 mmHg).
* Patients without current antihypertensive therapy.
* Patients on antihypertensive therapy, which can be stopped.
* 18 to 69 years of age.
* Male patients, or female patients without childbearing potential .

Exclusion Criteria:

* Patients with "very high added risk" according to 2007 Guidelines for the Management of Arterial Hypertension (Journal of Hypertension, 2007, 25:1105-1187), i.e. those with:
* grade III hypertension (mean sitting office SBP ≥180mmHg and/or mean sitting DBP≥110mmHg)
* history or presence of established cardiovascular or renal disease:
* Ischemic stroke, cerebral hemorrhage, transient ischemic attack
* Myocardial infarction, angina pectoris, coronary re-vascularization, heart failure
* Peripheral artery disease
* Diabetic nephropathy
* Known autoimmune disease.
* Severe allergy.
* Pregnancy or breastfeeding.
* Women in childbearing age that are not surgically sterilized.
* Patients with a history or current positive test for HIV infection, AIDS, or other immunosuppressive disorders; hepatitis B or C.
* Current diagnosis or history of malignancy.
* Presence of suspicious lymphadenopathy or splenomegaly on physical examination.
* Drug or alcohol abuse within the past 2 years.
* Presence or history of relevant cardiovascular, renal, hepatic, pulmonary, endocrine, autoimmune, neurological and psychiatric disease as judged by the investigator.
* Any current or past disease or conditions (physical or mental) that would, in the opinion of the investigator, interfere with the study procedures or interpretation of the study data (e.g. workers in the night shift).
* Previous participation in a clinical trial with a Qb based vaccine.
* Use of an investigational drug within 3 months before enrolment, or planned use during the whole study period.
* Possible dependency of the patient on sponsor and/or investigator.
* Planned active immunization 2 weeks before or 2 weeks after any study medication vaccination.
* Donation or loss >=400 mL of blood within 8 weeks prior to dosing or major surgery within past 2 months.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Adverse events: quality, quantity, severity | Throughout the study until week 48

SECONDARY OUTCOMES:
Change in daytime, nighttime and 24-hour ambulatory blood pressure from baseline | 24 hours
Titer of IgG specific for angiotensin II | Throughout the study untill week 48
Amount of RAS-Biomarkers (plasma renin concentration, angiotensin II, aldosterone) | 24 hours

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (2):
  - CRS Mannheim, Mannheim
  - CRS Mönchengladbach, Mönchengladbach
- Switzerland (4):
  - University Hospital Basel, Basel
  - Inselspital, Bern
  - Hopital Universitaire Geneve, Geneva
  - Med Zentrum Römerhof, Zurich